CLINICAL TRIAL: NCT07198841
Title: The Efficacy and Safety of IBI351 Plus Cetuximab β in Untreated, Locally Advanced or Metastatic Non-small Cell Lung Cancer With KRAS G12C Mutation: A Single-arm, Prospective, Multicenter Phase II Clinical Study
Brief Title: IBI351 Plus Cetuximab β in Untreated Advanced Non-small Cell Lung Cancer With KRAS G12C Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry); Mabpharm Limitied (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2506
Record Dates: First submitted 2025-08-27; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer (Non-Small Cell)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI351+ cetuximab β treatment (Experimental)
  Interventions: Drug: IBI351 combined with cetuximab β

INTERVENTIONS:
Drug: IBI351 combined with cetuximab β — Subjects will receive treatment with IBI351 plus cetuximab β, consisting of oral IBI351 administered at 600 mg twice daily (BID) either in a fasting or fed state, combined with intravenous infusion of cetuximab β injection dosed at 500 mg/m² (body surface area) every two weeks. Each treatment cycle spans two weeks. Therapy will continue until disease progression, unacceptable toxicity, or meeting other protocol-defined criteria for treatment discontinuation-whichever occurs first. Dose adjustments may be implemented throughout the study based on drug-related toxicities.

SUMMARY:
Study Design: a Phase II, single-arm, multicenter, prospective, interventional study.

Target Population: Subjects with previously untreated, locally advanced or metastatic non-small cell lung cancer (NSCLC) confirmed to harbor the KRAS G12C mutation.

Treatment Regimen: All enrolled subjects will receive IBI351 combined with cetuximab β injection. Treatment will continue until disease progression (as assessed by the investigator per RECIST 1.1 criteria) or the occurrence of intolerable toxicity.

Primary Endpoint: Objective Response Rate (ORR) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

Secondary Endpoints: Disease Control Rate (DCR), Time to Response (TTR), Progression-Free Survival (PFS), and Overall Survival (OS) , and safety.

ELIGIBILITY:
Inclusion Criteria

1. Voluntarily participate in the study and sign the informed consent form (ICF).
2. Male or female subjects aged ≥18 years and ≤75 years at the time of signing the ICF.
3. Life expectancy ≥ 3 months.
4. Histologically or cytologically confirmed unresectable locally advanced (Stage IIIB/IIIC), metastatic, or recurrent (Stage IV) non-small cell lung cancer (NSCLC), per the International Association for the Study of Lung Cancer (IASLC) and American Joint Committee on Cancer (AJCC) 8th edition TNM staging, and not candidates for curative concurrent chemoradiotherapy.
5. Documented KRAS G12C mutation confirmed by a written report from a certified laboratory.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.
7. No prior systemic anti-tumor therapy for locally advanced or metastatic non-squamous NSCLC. Subjects who received prior adjuvant therapy are eligible provided disease recurrence occurred ≥6 months after the last dose of adjuvant therapy or the last session of radical radiotherapy.
8. At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Lesions within a prior radiation field or after local therapy can be considered target lesions if documented progression is evident.
9. Adequate organ and bone marrow function, defined as:

1）Hematopoietic: Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L, platelet count ≥ 100 × 10⁹/L, hemoglobin ≥ 9 g/dL. No transfusion or treatment with granulocyte colony-stimulating factor (G-CSF), thrombopoietin, or erythropoietin within 14 days prior to hematology tests.

2）Hepatic: Total bilirubin (TBIL) < 1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 × ULN. For subjects with Gilbert's syndrome, TBIL < 2 × ULN is acceptable. For subjects with liver metastases, AST and ALT < 5.0 × ULN is required. If direct bilirubin (DBIL) suggests extrahepatic obstruction, TBIL < 3.0 × ULN is permitted.

3）Renal: Serum creatinine (Cr) ≤ 1.5 × ULN OR calculated creatinine clearance (CrCl) ≥ 60 mL/min (using the Cockcroft-Gault formula) if Cr > 1.5 × ULN.

4）Coagulation: Prothrombin time (PT) / activated partial thromboplastin time (APTT) < 1.5 × ULN and international normalized ratio (INR) < 1.5 or within the therapeutic range for subjects on anticoagulation therapy.

5）Magnesium: Serum magnesium within normal limits. 10. Toxicities from prior anti-tumor therapy must have resolved to baseline or ≤ Grade 1 (except for residual alopecia; neurotoxicity ≤ Grade 2 is acceptable). Subjects with prior immune-related endocrine adverse events (irAEs) from immunotherapy (e.g., hypothyroidism) that are asymptomatic and stably controlled with ongoing hormone replacement or physiologic doses of corticosteroids may be enrolled if the investigator judges that this will not affect study drug administration or safety assessment.

11. Female subjects of childbearing potential or male subjects with partners of childbearing potential must use effective contraception from signing the ICF until 6 months after the last dose of study drug. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days (inclusive) prior to the first dose. If a urine pregnancy test result is inconclusive, a serum pregnancy test is required.

Exclusion Criteria

1. Histologically or cytologically confirmed NSCLC with mixed small cell components or predominantly squamous cell carcinoma components.
2. Presence of EGFR sensitizing mutation, ALK rearrangement, ROS-1 fusion, or other genomic alterations for which NMPA-approved first-line NSCLC therapies exist.
3. Significant cardiovascular or cerebrovascular disease, including:

1）Clinically significant cardiovascular events within 6 months (e.g., myocardial infarction, angina, heart failure, severe arrhythmia) or history of angioplasty, stenting, or coronary artery bypass grafting.

2）Clinically significant prolongation of the QTcF interval (QTcF > 470 ms for females or > 450 ms for males).

3）Clinically significant cerebrovascular events within 3 months (e.g., cerebral hemorrhage, infarction).

4. Active central nervous system (CNS) metastases (e.g., brain or leptomeningeal metastases). Subjects with previously treated brain metastases may be eligible if they are asymptomatic for at least 7 days after completion of radiotherapy/local therapy without requiring steroids/anti-epileptics, OR off steroids/anti-epileptics for at least 7 days, AND judged by the investigator to have stable CNS disease.

5. Clinically significant interstitial lung disease (ILD), radiation pneumonitis, or drug-induced pneumonitis requiring treatment; active pulmonary tuberculosis; pneumoconiosis; Grade ≥2 pneumonitis of other etiologies; or severely impaired pulmonary function (FEV1 or DLCO or DLCO/VA <40% of predicted value).

6. Significant gastrointestinal disorders affecting drug absorption or swallowing (e.g., refractory hiccups, nausea, vomiting, severe peptic ulcer disease, liver cirrhosis, active GI bleeding).

7. Major active or chronic infections, including:

1. Active infection requiring systemic therapy.
2. Baseline positive HIV antibody (HIV-Ab); acute or chronic active hepatitis B (defined as HBsAg and/or HBcAb positive AND HBV-DNA > 2500 copies/mL or 500 IU/mL); or acute or chronic active hepatitis C (HCV antibody positive AND HCV-RNA above the lower limit of quantification).
3. Active pulmonary tuberculosis. 8. Symptomatic pleural, peritoneal, or pericardial effusions requiring repeated drainage.

9. Poorly controlled systemic diseases despite standard therapy (e.g., hypertension: systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg; diabetes).

10. History of other active malignancies within 2 years prior to study entry, except appropriately treated carcinoma in situ of the cervix, localized squamous cell carcinoma of the skin, basal cell carcinoma, prostate cancer not requiring treatment, ductal carcinoma in situ of the breast, and superficial non-muscle invasive urothelial carcinoma.

11. Prior treatment with any KRAS G12C inhibitor. 12. Prior treatment with cetuximab or its analogues. 13. Systemic treatment with Chinese herbal medicine with anti-tumor indications within 1 week prior to the first dose, OR systemic treatment with immunomodulatory drugs (including thymosin, interferon, interleukin; except for localized intrapleural use for effusion control) within 2 weeks prior to the first dose.

14. Therapeutic or palliative radiotherapy (except cranial radiotherapy) or local therapy within 14 days prior to the first study dose.

15. Any other anti-tumor therapy (chemotherapy, targeted therapy, immunotherapy, investigational drug/device) within 28 days or 5 half-lives (whichever is shorter) prior to the first study dose.

16. Major surgery within 28 days prior to study entry that could affect study drug administration or assessments (excluding diagnostic biopsy).

17. Use of known sensitive substrates of CYP2D6, CYP3A4, P-gp, or BCRP with a narrow therapeutic window within 14 days or 5 half-lives (whichever is longer) prior to the first study dose, unless agreed upon by both the investigator and sponsor.

18. Concurrent participation in another interventional clinical trial (participation in observational studies or the follow-up phase of an interventional study is permitted).

19. Use of immunosuppressive drugs within 4 weeks prior to the first study dose, excluding intranasal, inhaled, or topical corticosteroids; systemic corticosteroids at physiologic doses (≤10 mg/day prednisone or equivalent); or corticosteroids administered for prophylaxis of contrast media allergy.

20. Administration of live attenuated vaccines within 4 weeks prior to the first study dose or planned during the study period.

Note: Inactivated seasonal influenza vaccines administered >4 weeks prior are allowed; live attenuated influenza vaccines are not permitted.

21. Known or suspected autoimmune disease, or history of autoimmune disease within 2 years prior to screening (subjects with vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic therapy in the last 2 years, hypothyroidism managed only with hormone replacement, or type 1 diabetes managed only with insulin replacement are eligible).

22. Known history of primary immunodeficiency. 23. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

24. History of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolic event within 3 months prior to enrollment (implant port- or catheter-related thrombosis, or superficial venous thrombosis are not considered "severe").

25. Known hypersensitivity to any component of the study drug or its formulation.

26. Pregnant or breastfeeding women. 27. Any other condition that, in the investigator's judgment, would make the subject unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From the first dose of treatment to disease progression or death, whichever comes first, up to 2 years
  The proportion of patients achieving complete and partial response after treatment, measured according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression-Free Survival | From the first dose of treatment until the first documentation of disease progression or death from any cause, whichever occurs first (up to 2 years)
  Progression-free survival is defined as the time from first dose of treatment to the first documentation of disease progression or death from any cause, whichever occurs first. Disease progression will be assessed according to RECIST version 1.1 criteria
Time To Response | From the first dose to disease progression or death, whichever comes first, up to 2 years
  Time from the first administration of the drug to the first assessment by the investigator using RECIST 1.1 criteria as Complete Response or Partial Response
Disease Control Rate | From the first dose to disease progression or death, whichever comes first, up to 2 years
  Disease control rate is defined as the proportion of participants with complete response, partial response, and stable disease, as determined by RECIST v1.1 criteria
Overall Survival | From the first dose of treatment to death due to any reason, whichever comes first, up to 2 years
  The time from the first administration of treatment to death due to any reason
Adverse Events | From the first dose of treatment to disease progression or death (up to 2 years)
  Assessed by recording treatment-related adverse events and serious adverse events , graded according to the CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, Southern Medical University,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided